CLINICAL TRIAL: NCT01267929
Title: Effects of Mirror Neurons Stimulation on Motor Skill Rehabilitation in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thammasat University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Namfon Mahasup, Ph.D.candidate, Postgraduate Studied Program, faculty of Medicine, Thammasat University, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTU-P-1-71/51
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Children With Spastic Diplegia, Between the Ages of 2 to 10 Years; Gross Motor Function Classification System (GMFCS) Level I,II and III
Keywords: Children with cerebral palsy; Gross Motor Function Measure; Imitative learning; Mirror neuron; Action observation; Conventional physical therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The mirror neurons stimulation based VCD program (Experimental): The children receive the mirror neurons stimulation based VCD program and practice at home three times a day for six months. The mirror neurons stimulation based VCD program that contained four volumes. The first volume includes activities activities for improving balance in sitting position. The second volume includes activities of sitting to standing. The third volume includes activities for improving balance in standing position. The last one includes activities of sideway walking. The running time of each volume is 30 minutes. The children had been practicing for two weeks per volume. Their parents were trained for practicing their children by VCD program at home and were asked to complete daily record of children's activities. The children were scheduled to meet a pediatric physical therapist once a week to monitor possible side effects.
  Interventions: Procedure: The mirror neurons stimulation based VCD program
- The conventional physical therapy (Active Comparator): The children receive manual physical therapy regularly at the hospital once a week for first two months and twice a month for last four months. The conventional physical therapy technique in this study derive from the manual technique including the Bobath concept, stretching exercise and functional training for 30-45 minutes at a time.
  Interventions: Procedure: The conventional physical therapy

INTERVENTIONS:
Procedure: The mirror neurons stimulation based VCD program — The children receive the mirror neurons stimulation based VCD program and practice at home three times a day for six months.
  Arms: The mirror neurons stimulation based VCD program
Procedure: The conventional physical therapy — The children were randomly assigned to receive the conventional physical therapy for six months. Both experimental and control groups were measured their motor functions with GMFM-66 by an independent pediatric physical therapist who was blinded for treatment allocation at entry, the second month and the sixth month.
  Arms: The conventional physical therapy

SUMMARY:
This study aimed to develop Video Compact Disc (VCD) program that applying the concept of imitative learning with mirror neurons stimulation on standard rehabilitation technique in children with cerebral palsy. The author will also examine effectiveness of the program by compare the motor function measured by the gross motor function measure (GMFM-66) between conventional physical therapy and the mirror neurons stimulation based VCD program for six months.

DETAILED DESCRIPTION:
A randomized controlled trial was performed with thirty children with cerebral palsy recruited from Thammasat University Hospital and Rajanukul institute. Informed consent was obtained from the participants' parents before participation in this study. The participants were randomly assigned according to the randomization list to receive either the mirror neurons stimulation based VCD program and practice at home or conventional physical therapy for six months. The participants in the experiment group received the mirror neurons stimulation based VCD program and practice at home three times a day for six months. Concerning the control group, the participants received conventional physical therapy regularly at the hospital once a week for first two months and twice a month for last four months. Both experimental and control groups were measured their motor functions with gross motor function measure (GMFM-66).

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy aged between 2-10 years old
* GMFCS level of one to three
* Able to verbal instruction
* Sitting are performed without assistance
* Standing and walking are performed with adult assistance
* No severe limitation of joint movement

Exclusion Criteria:

* The children were received orthopedic intervention or botulinum toxin injection within 6 months
* Seizure
* Other conditions that prevent children from participate in research project
* Severe visual and hearing deficits

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-09; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Assoc.Prof.Paskorn Sritipsukho, MD, Study Director — Thailand:Faculty of Medicine Thammasat University
Locations (1):
- Department of Physical therapy, Faculty of Allied Health Sciences Thammasat University, Pathum Thani, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The children were recruited from Thammasat University hospital and Rajanukul institute. Study period was two years which started from September 2009 to October 2011.
Pre-assignment Details: Thirty two children were assessed for their eligibility to participate in the study. One were excluded for failing to meet the inclusion criteria. One parent of a child refused to participate in the study.
Groups:
- The Mirror Neurons Stimulation Based VCD Program: The children receive the mirror neurons stimulation based Video Compact Disc (VCD) program and practice at home three times a day for six months. The mirror neurons stimulation based VCD program that contained four volumes. The first volume includes activities activities for improving balance in sitting position. The second volume includes activities of sitting to standing. The third volume includes activities for improving balance in standing position. The last one includes activities of sideway walking. The running time of each volume is 30 minutes. The children had been practicing for two weeks per volume. Their parents were trained for practicing their children by VCD program at home and were asked to complete daily record of children's activities. The children were scheduled to meet a pediatric physical therapist once a week to monitor possible side effects.
Period: Overall Study
Arm/Group | The Mirror Neurons Stimulation Based VCD Program | The Conventional Physical Therapy
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Mirror Neurons Stimulation Based VCD Program | The Conventional Physical Therapy | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] — The average age of each group
  years | 6.2 (2.2) | 5.5 (2.2) | 5.9 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants] — The number of males and females of each group
  Participants
    Female | 6 | 5 | 11
    Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  Thailand | 15 | 15 | 30
Baseline Gross Motor Function Measure (GMFM-66) score [Mean (Standard Deviation); unit: Scores] — The mean total score of GMFM-66 of each group at entry. The GMFM-66 contains five dimensions of motor measure including lying/rolling (4 items), sitting (15 items), crawling/kneeling (10 items), standing (13 items), and walking/running/jumping (24 items). The GMFM-66 are scored on a 4-point ordinal scale 0=does not initiate, 1=initiates < 10% of activity,2=partially completes 10% to < 100% of activity,3=completes activity). The scores were converted to a continuous scale by using the Winsteps Rasch Software. GMFM-66 score less than 30 that are considered low gross motor skills.
  Scores | 44.8 (14.0) | 49.4 (13.1) | 47.1 (13.5)

OUTCOME MEASURES:

1. Primary Outcome: The Gross Motor Function Measure (GMFM-66) Score at Entry, the Second and the Sixth Month.
Description: The mean total score of GMFM-66 of each group at entry, the second and the sixth month. The GMFM-66 contains five dimensions of motor measure including lying/rolling (4 items), sitting (15 items), crawling/kneeling (10 items), standing (13 items), and walking/running/jumping (24 items). The GMFM-66 are scored on a 4-point ordinal scale 0=does not initiate, 1=initiates < 10% of activity,2=partially completes 10% to < 100% of activity,3=completes activity). The scores were converted to a continuous scale by using the Winsteps Rasch Software.The GMFM-66 score is an interval-level measure of function where subjects are placed on an ability continuum ranging from 0 (low motor ability) to 100 (high motor ability). GMFM-66 score less than 30 that are considered low gross motor skills.
Time Frame: Base line, two months and six months
Population: A total of 30 children with cerebral palsy was followed and completed the study.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | The Mirror Neurons Stimulation Based VCD Program | The Conventional Physical Therapy
Number analyzed (Participants) | 15 | 15
Scores on a scale
  The mean score of GMFM-66 at the entry | 44.8 (14.0) [37.4 to 52.1] | 49.4 (13.1) [42.5 to 56.3]
  The mean score of GMFM-66 at the second month | 54.7 (14.5) [25.2 to 70.2] | 57.5 (16.2) [31.3 to 80.4]
  The mean score of GMFM-66 at the sixth month | 57.8 (13.9) [50.4 to 65.1] | 63.2 (16.8) [54.3 to 72.1]
Statistical Analysis 1: Comparison: The Mirror Neurons Stimulation Based VCD Program vs The Conventional Physical Therapy; A sample size of 30 children, 15 for each group, was needed to obtain 80% power at 0.05 level of significance (two-sided) to test that the successful event rate (increasing GMFM scores at least 30% from baseline at the end of 2 months) in experimental group and control group of 0.3 and 0.8 respectively. The mean changes of GMFM total scores in the experimental group at the second month compared to those in the control group after adjusted for the baseline level; Test type: Superiority or Other; p = 0.34, ANCOVA — Statistical analysis was conducted using STATA. Analysis of Covariance (ANCOVA) was used to compare mean score of GMFM at the second month between two groups; Mean Difference (Final Values) = 2.1, 95% CI 2-sided [-2.3 to 6.5], Standard Error of Mean 2.14
Statistical Analysis 2: Comparison: The Mirror Neurons Stimulation Based VCD Program vs The Conventional Physical Therapy; A sample size of 30 children, 15 for each group, was needed to obtain 80% power at 0.05 level of significance (two-sided) to test that the successful event rate (increasing GMFM scores at least 30% from baseline at the end of 2 months) in experimental group and control group of 0.3 and 0.8 respectively. The mean changes of GMFM total scores in the experimental group at the sixth month compared to those in the control group after adjusted for the baseline level; Test type: Superiority or Other; p = 0.78, ANCOVA — Statistical analysis was conducted using STATA. Analysis of Covariance (ANCOVA) was used to compare mean score of GMFM at the sixth month between two groups; Mean Difference (Net) = -0.7, 95% CI 2-sided [-6.3 to 4.7], Standard Error of Mean 2.7

ADVERSE EVENTS:
Arm/Group | The Mirror Neurons Stimulation Based VCD Program | The Conventional Physical Therapy
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
This Video Compact Disc (VCD) program was applicable for children with cerebral palsy with spastic diplegia who had high GMFCS level (1-3). Generalized the results to children with other types of cerebral palsy with different severity are limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No